CLINICAL TRIAL: NCT00243399
Title: A Pilot Trial of Oxandrolone for the Treatment of Bone Marrow Aplasia in Patients With Fanconi Anemia
Brief Title: Oxandrolone for the Treatment of Bone Marrow Aplasia in Fanconi Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Franklin O. Smith, Cincinnati Children's Hospital Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2539; FD-R-002539-01
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia; FA
MeSH Terms: conditions — Fanconi Anemia | interventions — Oxandrolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxandrolone (Experimental)
  Interventions: Drug: Oxandrolone

INTERVENTIONS:
Drug: Oxandrolone — Subjects will be started on a dose of oxandrolone 0.04 mg/kg/day orally, once/day. After 16 weeks, patients will be assessed for hematologic improvement. If this criteria is not met after 16 weeks, the dose will be escalated to 0.08 mg/kg/day. If no improvement is noted after 16 weeks on the escalated dose, oxandrolone therapy will be discontinued.
  Other Names: Oxandrin

SUMMARY:
The purpose of this study is to evaluate the safety of the drug oxandrolone (a type of androgen steroid) in patients with Fanconi anemia (FA), and to determine if this drug can help in the treatment of bone marrow failure in these patients. Androgen steroids are male hormones that can stimulate the production of red blood cells (the cells which carry oxygen in the blood) and platelets (cells that help blood clot).

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the safety of the drug oxandrolone in patients with Fanconi anemia (FA), and secondarily to determine if this drug can help in the treatment of bone marrow failure in these patients. It is hoped that oxandrolone will have less side effects than oxymetholone, the androgen used most frequently in the short-term treatment of bone marrow failure in FA patients. Subjects will be enrolled for approximately 18 to 30 months (12 - 24 months of treatment and 6 months additional monitoring). The oxandrolone starting dose is 0.04mg/kg/day. Study monitoring includes weekly complete blood counts, monthly serum chemistry labs, quarterly physical examinations including virilization exams and liver ultrasounds. Semi-annually, hand radiographs are obtained for bone maturation and behavioral assessments are conducted to detect any aggressive behavior or mood changes. If no improvement n the subject's blood counts are noted after 4 months of therapy, the dose will be increased to 0.08mg/kg/day for a period of 4 more months. If no improvement is noted after a total of eight months, oxandrolone will be discontinued. If the blood counts show improvement, then the drug will continue for a minimum of twelve months. Subjects may remain on study and receive a total of 24 months of therapy if they have a response in their blood counts without unacceptable side effects. Post-treatment monitoring includes blood work and ultrasound every three months, and hand radiograph at six months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with Fanconi anemia that is documented by a positive test for increased chromosomal breakage with mitomycin C or diepoxybutane.
2. At least the following peripheral blood cytopenias: (without transfusion) Absolute neutrophil count < 500/mm3 or Platelet count < 30,000/mm3 or Hemoglobin < 8.0 gm/dl
3. Negative pregnancy test by hCG testing, if of child-bearing potential.
4. Agreement to use a medically approved form of birth control, if of child-bearing potential.
5. Signed informed consent by the patient or legally authorized representative.
6. Patients must be 14 kg.
7. Male patients will be included until the time of puberty. With the onset of puberty, they will be included until the testosterone levels reach 100 ng/dl at which time they will be excluded from the study.

Exclusion Criteria:

1. Malignancy
2. Concurrent enrollment in any other study using an investigational drug.
3. Concurrent use of anticoagulants.
4. Use of androgen therapy within last three months.
5. Patients with severe liver disease as defined by SGOT or SGPT greater than or equal to 2.5x the upper limit of normal or total bilirubin greater than or equal to 1.5x the upper limit of normal.
6. Patients with renal disease as defined by serum creatinine greater than or equal to 1.5 x the upper limit of normal for age.
7. Patients less than 14 kg.
8. Patients who have failed previous therapy with oxymetholone.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-07; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Toxicity associated with oxandrolone therapy in patients with Fanconi Anemia | One year

SECONDARY OUTCOMES:
Hematologic response rate in Fanconi Anemia patients receiving oxandrolone therapy | One year

CONTACTS AND LOCATIONS:
Overall Officials: Franklin O Smith, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States